CLINICAL TRIAL: NCT05277038
Title: Clonidine is Better Than Zopiclone for Insomnia Treatment in Chronic Pain Patients
Status: Completed | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnaesth 2021 ClonZop
Record Dates: First submitted 2022-01-25; First posted 2022-03-14 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-03

CONDITIONS: Insomnia Chronic; Pain, Chronic
Keywords: sedative; hypnotic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain | interventions — Clonidine; Tablets; zopiclone

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clonidine vs Zopiclone for insomnia: Consecutive adult patients who underwent pain management at a Canadian pain clinic. The patients were subsequently prescribed and provided zopiclone 3.75mg tablet (1-2 tablets per dose), and clonidine 0.1mg tablet (1-2 tablets per dose). They were advised to take either clonidine or zopiclone on alternate nights. For each medication, they alternated the doses of 1 tablet or 2 tablets at subsequent nightly administrations. The four possible medication doses were zopiclone 3.75mg, zopiclone 7.5mg, clonidine 0.1mg, and clonidine 0.2mg; as shown on the sleep diary in Figure 1. The recommended orders of treatment were zopiclone 7.5mg, clonidine 0.1mg, zopiclone 3.75mg, clonidine 0.2mg; or clonidine 0.2mg, zopiclone 3.75mg, clonidine 0.1mg, zopiclone 7.5mg. Each patient participated in the study treatment and completed the sleep diary for 3 continuous weeks. Therefore, each of the four medication doses was used five times by each patient.
  Interventions: Drug: Clonidine 0.1mg pill; Drug: Clonidine 0.2mg pill; Drug: Zopiclone 3.75mg pill; Drug: Zopiclone 7.5mg pill

INTERVENTIONS:
Drug: Clonidine 0.1mg pill — Routine prescription for insomnia
  Other Names: Clonidine 0.1mg tablet
Drug: Clonidine 0.2mg pill — Routine prescription for insomnia
  Other Names: Clonidine 0.2mg tablet
Drug: Zopiclone 3.75mg pill — Routine prescription for insomnia
  Other Names: Zopiclone 3.75mg tablet
Drug: Zopiclone 7.5mg pill — Routine prescription for insomnia
  Other Names: Zopiclone 7.5mg tablet

SUMMARY:
A prospective observational crossover study of 160 consenting adult patients who underwent pain management. For insomnia treatment, each patient ingested different prescribed doses of Zopiclone or Clonidine on alternate nights. Each patient used a special validated sleep diary to collect data including pain score, sleep scores, sleep duration, sleep medication dose, and adverse effects. Each patient completed the diary for 3 continuous weeks. Pain was measured using the numeric pain rating scale. Sleep score was measured using the Likert sleep scale. A change in the pain or sleep scores by 2-points was considered significant.

DETAILED DESCRIPTION:
Objectives: Chronic pain is associated with insomnia. The objective of this clinical study is to compare the efficacy and safety of different prescribed doses of Zopiclone and Clonidine; for the management of insomnia in patients with chronic pain.

Methods: A prospective observational crossover study of 160 consenting adult patients who underwent pain management. For insomnia treatment, each patient ingested different prescribed doses of Zopiclone or Clonidine on alternate nights. Each patient used a special validated sleep diary to collect data including pain score, sleep scores, sleep duration, sleep medication dose, and adverse effects. Each patient completed the diary for 3 continuous weeks. Pain was measured using the numeric pain rating scale. Sleep score was measured using the Likert sleep scale. A change in the pain or sleep scores by 2-points was considered significant. Data were analyzed with IBM® SPSS® Statistics 25 (IBM Corp, Armonk, NY); using Student's t-test, ANOVA, Pearson Chi-square test, and regression analysis. P-value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients
* good treatment compliance
* severe chronic insomnia
* failure of non-pharmacologic sleep therapy
* regular zopiclone therapy for 3 months or more
* regular sleep diary
* regular pain diary
* informed consent for diary review
* consent for clinical record quality assurance review.

Exclusion Criteria:

* obstructive sleep apnoea
* body mass index (BMI) ≥40
* organ insufficiency
* cognitive disorder
* inability to provide consent
* major neuropsychiatric disorder
* unreliable diary
* cannabis use
* regular alcohol intake
* stimulant use
* substance abuse
* poor treatment compliance
* high dose opioid
* gabapentinoid use
* sedative use
* mild insomina
* irregular zopiclone intake
* regular zopiclone therapy for less than 3 months
* previous adverse/allergic reactions to clonidine or zopiclone.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of consecutive adult patients who underwent pain management at a Canadian pain clinic
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Sleep quality score, objective measurement using the validated Likert sleep scale | 3 weeks
  Sleep quality score, using the Likert sleep scale of 0 to 10, low scores indicate poor sleep, high scores indicate better sleep

SECONDARY OUTCOMES:
Pain score, objective measurement using the validated Numeric Pain Rating scale | 3 weeks
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD, FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lader M. Zopiclone: is there any dependence and abuse potential? J Neurol. 1997 Apr;244(4 Suppl 1):S18-22. doi: 10.1007/BF03160567. PMID 9112585